CLINICAL TRIAL: NCT07043439
Title: Comparison of the Immediate Effects of Mobilization and Manipulation Versus Sham Manipulation on Plantar Pressure in Patients With Hallux Valgus
Acronym: HALLPRESS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SEFA HAKTAN HATIK (Other)
Responsible Party: Sponsor-Investigator, SEFA HAKTAN HATIK, Asst. Professor, Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMT0009
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Hallux Valgus; Foot Deformities; Musculoskeletal Manipulations; Plantar Pressure; Manuel Therapy; Chiropractic
Keywords: Hallux Valgus; First Metatarsal Mobilization; HVLA Manipulation; Sham Manipulation; Plantar Pressure Analysis; Pedobarography; Manual Therapy; Chiropractic Mobilization; Pain; Quality of Life
MeSH Terms: conditions — Hallux Valgus; Foot Deformities; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study will employ single masking. The outcomes assessor will be blinded to the group allocation of the participants (intervention vs. sham). Participants and therapists will not be blinded due to the nature of manual interventions, which require active therapist involvement and differ in technique between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization and Manipulation Group (MMG) (Experimental): Participants in this group underwent high-velocity, low-amplitude (HVLA) chiropractic manipulation of the first metatarsophalangeal (MTP) joint by an experienced physical therapist, followed by grade 3 accessory mobilization.
  Participants were placed in the prone (face-down) position during the procedure, and the foot was stabilized in a neutral position.
  Manipulation: The therapist stabilized the first metatarsal bone with one hand while applying a quick, short traction force to the proximal phalanx of the first toe with the other hand.
  Mobilization: Following manipulation, grade 3 rhythmic oscillations were applied to the same joint in accordance with the Maitland technique to increase joint play.
  The entire procedure was completed in a single session, with evaluations conducted immediately before and after the intervention.
  Interventions: Other: Mobilization; Other: High-Velocity Low-Amplitude (HVLA) Manipulation
- Control Group (CG) (Sham Comparator): The control group individuals underwent sham manipulation in the same position (prone and neutral foot) and for the same duration. During the sham application, the therapist assumed the manipulation position, placed his hands on the first metatarsal, and created the impression that the application was being performed. However, no traction, pushing, mobilization, or high-speed movement was applied during this process.
  This application was performed in a way that would make the participant believe they were receiving treatment, but without creating any biomechanical or neurophysiological effects.
  Since the purpose of the sham group was to control for the placebo effect, evaluations were also conducted on the individuals in this group before and immediately after the application.
  For ethical reasons, the real treatment protocol was also applied to these participants after the evaluations.
  Interventions: Other: Sham Manipulation

INTERVENTIONS:
Other: Mobilization — Participants receiving this intervention will undergo Grade 3 joint mobilization targeting the first metatarsophalangeal (1st MTP) joint. The technique will be administered by a licensed physiotherapist with the participant lying in the prone position and the foot in a neutral position.
  Mobilization will be performed according to the Maitland concept, which defines Grade 3 as large-amplitude, rhythmic oscillatory movements applied within the range of motion but up to the limit of tissue resistance, without entering the paraphysiological space.
  The goal of this technique will be to increase joint play and mobility, reduce stiffness, and potentially improve biomechanical alignment. The mobilization will last approximately 5 minutes, and outcome measures will be collected before and immediately after the session.
  Arms: Mobilization and Manipulation Group (MMG)
Other: High-Velocity Low-Amplitude (HVLA) Manipulation — This intervention will involve the application of a high-velocity, low-amplitude (HVLA) thrust manipulation to the first metatarsophalangeal (1st MTP) joint. A licensed physiotherapist will perform the procedure with the participant positioned prone and the foot placed in a neutral alignment.
  The therapist will stabilize the 1st metatarsal bone with one hand and apply a quick, controlled thrust to the proximal phalanx of the hallux in a dorsal direction using the other hand. The technique will be delivered with minimal amplitude and maximal speed, aiming to restore joint motion, reduce soft tissue tension, and stimulate neuromechanical reflexes.
  The manipulation procedure will take approximately 2-3 minutes, including setup and execution. Pre- and post-intervention outcome measures will be used to assess its immediate effects.
  Arms: Mobilization and Manipulation Group (MMG)
Other: Sham Manipulation — Participants in the control group will receive a sham (placebo) intervention designed to mimic the real treatment in setup and duration, without applying any therapeutic mechanical stimulus. The sham procedure will be conducted by the same physiotherapist with participants lying prone and their foot in a neutral position.
  The physiotherapist will place their hands around the 1st MTP joint as if a manipulation were to be performed and will maintain static contact for the same duration as in the experimental group. However, no thrust, traction, or mobilization force will be applied.
  The sham intervention will also last approximately 10 minutes, ensuring consistency across groups. All assessments will be conducted immediately before and after the intervention to evaluate potential placebo effects.
  Arms: Control Group (CG)

SUMMARY:
The aim of this study is to examine the immediate effects of mobilization and manipulation versus sham manipulation on plantar pressure, quality of life, and pain in patients with hallux valgus. Participants will be assessed using a sociodemographic data form, the Manchester-Oxford Foot Questionnaire (MOXFQ), the Manchester Scale, goniometric measurements, the Multidimensional Nil Hallux Valgus Scale, the SF-36 Health Survey, the Numeric Pain Rating Scale (NPRS), and plantar pressure analysis via a pedobarographic device. The study will be conducted on a total of 60 feet, with 30 feet assigned to the manipulation group and 30 feet to the sham manipulation group.

DETAILED DESCRIPTION:
This is a single-center interventional study to be conducted at Diagenics R&D Technology Health Import and Export Co. Ltd., aiming to explore the biomechanical impact of manual therapy techniques in individuals with hallux valgus. The study focuses on the immediate effects of first metatarsal mobilization and high-velocity, low-amplitude (HVLA) chiropractic manipulation, compared to a sham procedure, on plantar pressure distribution.

In the intervention group, participants will receive both grade 3 mobilization and HVLA manipulation targeted at the first metatarsophalangeal joint. The procedures will be carried out by a physiotherapist with the participant in a prone position and the foot held in neutral alignment.

The control group will receive a sham manipulation applied under identical positioning and handling conditions, but without therapeutic force or joint cavitation. This approach is designed to mimic the procedure while avoiding any real biomechanical impact. To eliminate ethical concerns regarding withholding effective treatment, participants in the control group will be offered the actual intervention after all immediate post-intervention data are collected.

All interventions and assessments will be conducted on a single day. Pre- and post-intervention plantar pressure data will be captured using a pedobarographic system. Pain intensity, joint angles, and other self-reported outcomes will be recorded using validated tools, but their details are provided in the corresponding modules.

The study's novelty lies in its integration of pedobarography for objective quantification of plantar pressure changes following isolated manual interventions, which may offer new insight into the acute mechanical responses of the foot in hallux valgus cases.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age
* Volunteer to participate in the study
* Have hallux valgus (those with a hallux valgus angle greater than 15 and a Manchester Scale score of B or higher)

Exclusion Criteria:

* Having undergone surgery on the foot or ankle area within the last 6 months
* Having any neurological or psychiatric problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
Pedobarographic Analysis | Baseline and immediately after the intervention (within the same session)
  Dynamic plantar pressure distribution will be measured using a computerized pedobarography system. Key parameters will include peak pressure, pressure-time integral, and contact area under specific foot regions (e.g., forefoot, hallux). The goal is to evaluate the immediate biomechanical effects of the intervention.
Goniometric Measurement of 1st MTP Joint Range of Motion | Baseline and immediately after the intervention (within the same session)
  Passive range of motion (flexion and extension) of the first metatarsophalangeal joint will be assessed using a standard goniometer. Measurements will be taken to detect acute changes in joint mobility after intervention.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline and immediately after the intervention (within the same session)
  Participants will rate their perceived pain level during weight-bearing using a numeric scale from 0 (no pain) to 10 (worst possible pain). This will help assess any acute analgesic effects of the intervention.
Manchester-Oxford Foot Questionnaire (MOXFQ) | Baseline and immediately after the intervention
  A validated self-reported questionnaire assessing foot-related pain, walking/standing difficulties, and social interaction limitations. Although designed for chronic use, it will be used to observe short-term perceptual changes.
Manchester Scale for Hallux Valgus Severity | Baseline and immediately after the intervention
  A visual grading scale used to classify the severity of hallux valgus deformity. While structural changes are not expected in the short term, it will be used for documentation and potential perceptual variation.
Multidimensional Nil Hallux Valgus Scale | Baseline and immediately after the intervention
  A multidimensional scale evaluating hallux valgus symptoms, appearance, shoe fit, and function. Will be used to assess changes in self-perception and functional symptoms.
SF-36 Short Form Health Survey | Baseline and immediately after the intervention
  A general health-related quality of life questionnaire consisting of 8 domains. Although designed for long-term monitoring, it will be applied to explore immediate changes in perceived well-being.

CONTACTS AND LOCATIONS:
Overall Officials: SEFA H HATIK, Asst. Prof., Principal Investigator — Sinop University
Locations (1):
- Sinop University, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No